CLINICAL TRIAL: NCT03603626
Title: Effect of Preemptive Pregabalin for Post-operative Pain Relief in Myringoplasty
Brief Title: Preemptive Pregabalin in Myringoplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the article is not a clinical trial but is a hospital based randomized comparative study. This was inadvertently uploaded.
Sponsor: Dhulikhel Hospital (Other)
Collaborators: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Ashish Dhakal, Lecturer, Department of Otolaryngology Head and Neck Surgery, Dhulikhel Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/18
Record Dates: First submitted 2018-07-07; First posted 2018-07-27 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Post-operative Analgesia; CSOM - Chronic Suppurative Otitis Media
Keywords: Endoscopic ear surgery; Myringoplasty; Pregabalin; Preemptive analgesia
MeSH Terms: interventions — Pregabalin; Folic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preemptive pregabalin (Experimental)
  Interventions: Drug: Pregabalin 150mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Pregabalin 150mg — Preemptive pregabalin 150 mg administered 1 hour before surgery
  Arms: Preemptive pregabalin
Drug: Placebo oral capsule — Placebo administered 1 hour before surgery
  Other Names: Vitamin B capsule
  Arms: Placebo

SUMMARY:
The aim of this study was to investigate the effect of preemptive pregabalin on post-operative pain reduction after myringoplasty.

DETAILED DESCRIPTION:
Patient were randomly assigned to one of two groups with 30 participants each by lottery method. Pregabalin group received capsule Pregabalin 150mg and Placebo group were given Vitamin B capsule 1 hour prior to surgery.

All patients underwent endoscopic myringoplasty with tragal cartilage and perichondrium graft. Surgical procedure was done under local anesthesia. 5ml of 2% xylocaine with 1:2,00,000 adrenalin was infiltrated in the four quadrants of external ear canal and on tragus. Around 2cm incision was given on canal surface of tragus and around 2cm x 1.5cm cartilage- perichondrium graft was obtained. The skin was closed with 4/0 prolene interrupted suture. Using rigid Hopkins II 0-degree endoscope (Karl Storz) with 4-millimeter diameter and 18 centimeters in length, margin of perforation was refreshed. Gelatin sponge was kept in the middle ear and cartilage perichondrium graft placed. Canal was then packed with gelatin soaked in ciprofloxacin ear drops followed by ribbon pack medicated with soframycin. Small dressing was applied over it.

Post-operative pain severity was assessed with VAS scale at 6, 12, 24, 48 hours. Rescue analgesia is given with Injection Ketorolac (30mg IV) or Tab Flexon (Ibuprofen 400mg + Paracetamol 500mg) whenever the patient required.

ELIGIBILITY:
Inclusion Criteria:

* Cases of Chronic suppurative otitis media (CSOM) inactive planned for endoscopic myringoplasty under local anesthesia,
* Age >= 18 years
* either sex.

Exclusion Criteria:

* Revision cases,
* Pregnancy or breastfeeding,
* Known or suspected sensitivity or contraindication to pregabalin,
* Patient using medication for chronic pain,
* History of seizure disorder,
* Mental retardation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
This study is constructed to determine whether the use of preemptive single dose oral pregabalin would decrease post-operative pain in patient undergoing myringoplasty. | At 6, 12, 24, 48 hours in postoperative period
  Post-operative pain severity was assessed with Visual Analogue Scale (VAS). It's a 10cm scale in which 0 represents no pain at all and 10 represents the worst pain imaginable. VAS score was compared between 2 groups at 6, 12, 24, 48 hrs post-operative period. This would show if there is any change in pain score between groups using pregabalin or placebo in the given time frame.

CONTACTS AND LOCATIONS:
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Kavre, Nepal